CLINICAL TRIAL: NCT01721018
Title: A Phase I/IIa Study of the Safety, Tolerability and Biological Effect of Single and Repeat Administration of the Selectively Replication-competent Herpes Simplex Virus HSV1716 Into the Tumor-bearing Pleural Cavity (Intrapleural) in Patients With Inoperable Malignant Pleural Mesothelioma.
Brief Title: Intrapleural Administration of HSV1716 to Treat Patients With Malignant Pleural Mesothelioma.
Acronym: 1716-12
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Virttu Biologics Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1716-12
Record Dates: First submitted 2012-10-22; First posted 2012-11-02 (Estimated); Last update posted 2017-06-09 (Actual); Status verified 2017-06

CONDITIONS: Malignant Pleural Mesothelioma
Keywords: Oncolytic virus; HSV1716; Mesothelioma; MPM; Woll; Sheffield; Weston Park; Virttu; Crusade
MeSH Terms: conditions — Mesothelioma, Malignant; Mesothelioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HSV1716 (Experimental): Single Arm Phase I/II study of intra-pleural HSV1716 administration.
  Interventions: Biological: HSV1716 Intra-pleural delivery

INTERVENTIONS:
Biological: HSV1716 Intra-pleural delivery
  Other Names: Seprehvir

SUMMARY:
HSV1716, an oncolytic virus, is a mutant herpes simplex virus (HSV) type I, deleted in the RL1 gene which encodes the protein ICP34.5.

Malignant mesothelioma is an aggressive, asbestos-related tumour of the pleural and peritoneal cavities. It is a rare cancer which occurs in individuals who have been exposed to asbestos, although it typically occurs decades after exposure (10-40 years later). Malignant pleural mesothelioma forms plaques that are distributed on the surface of the pleural space in the lung. Approximately 30% of patients require an indwelling pleural catheter for drainage of pleural effusions. In this patient group, the indwelling catheter may be used to facilitate loco-regional delivery of HSV1716 to the pleural space.

This study seeks to evaluate the safety and biological effects of single and multiple administrations of HSV1716 in the treatment of malignant pleural mesothelioma.

DETAILED DESCRIPTION:
The study will be conducted in two parts. PART A is a single centre, single dose design, open label. Patients with inoperable malignant pleural mesothelioma will receive a single dose of HSV1716 by intrapleural administration. Delivery will be by direct administration via an indwelling catheter into the pleural cavity. PART B is a single centre, repeat dose design, open label. Two groups of three patients with inoperable malignant pleural mesothelioma will receive 2 (group 1) or 4 (group 2) single doses of HSV1716 at weekly intervals. Administration will be via an indwelling catheter into the pleural cavity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven malignant pleural mesothelioma
* Patients with disease which is not amenable to potentially curative resection
* Patients with pleural effusions and/or 'trapped lung' who (i) have an existing indwelling pleural catheter for draining of excess pleural fluid or (ii) who require the insertion of an indwelling pleural catheter to drain excess pleural fluid
* Patients with a performance status ≤ 2 (ECOG)
* Age of ≥ 18 years (at screening)
* Ability to give written informed consent as evidenced by signature on the patient consent form, to communicate well with the investigator and to comply with the expectations of the study

Exclusion Criteria:

* Patients likely to require palliative radio- or chemotherapy within 30 days
* Any evidence of uncontrolled cardiac or respiratory disease that would be a contra-indication for virus administration
* Any other serious medical or psychiatric disorder that would be a contra-indication for virus administration
* Acute active infection of any kind or other severe systemic disease or medical or surgical condition that is deemed significant by the principal investigator
* Patients with immunosuppressive disorders or on systemic steroids > 5mg prednisolone/day
* Pregnancy: women of childbearing potential not taking adequate contraception, and women who are breast feeding
* Previous treatment with investigational viral therapy products
* Administration of any unlicensed or investigational product within 8 weeks of entry to the study
* No prior or concurrent malignancy within 5 years other than basal cell carcinoma of the skin or in situ neoplasia of the cervix uteri
* Inadequate haematological function as defined by:

Haemoglobin (Hb) < 10g/dl, Neutrophil Count < 1.5 x 10e9/l, Platelets < 100 x 10e9/l

* Deranged liver function tests: serum bilirubin ≥ 1.5 x upper limit of normal reference range for laboratory; transaminases ≥ 5 x upper limit of normal reference range
* Patients with inadequate renal function: serum creatinine ≥ 1.5 x upper limit of reference range for laboratory
* Patients whose indwelling catheter is not of the type approved by the sponsor for use in the study
* Outwith any of the inclusion criteria above or considered unsuitable for entry into the study in any other way at the discretion of the principal investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-10; Primary Completion 2016-11-14 (Actual); Study Completion 2016-11-14 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of HSV1716 given by single and repeat intrapleural administration in patients with inoperable malignant pleural mesothelioma. | Dose limiting toxicities will be assessed at 28 days after last injection of HSV1716.

SECONDARY OUTCOMES:
Obtain evidence of HSV1716 replication and lysis of malignant pleural mesothelioma cells through analysis of pleural fluid and serum samples for evidence of cell death and/or HSV1716 replication and/or changes in appropriate biomarkers. | Samples will be collected at each outpatient visit up to day 29 (Part A), or day 50 (Part B).

OTHER OUTCOMES:
Tumour measurement as recorded by CT scans and assessed using the modified Response Criteria in Solid Tumors (RECIST) for MPM. | CT scans at Baseline, day 29 and day 57.

CONTACTS AND LOCATIONS:
Overall Officials: Penella J Woll, MB BS PhD FRCP, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust, Weston Park Hospital, Sheffield, S10 2SJ, UK
Locations (2):
- United Kingdom (2):
  - Weston Park Hospital, Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, South Yorkshire
  - Queen Elizabeth Univeristy Hospital, NHS Greater Glasgow & Clyde Health Board, Glasgow